CLINICAL TRIAL: NCT00993707
Title: A Phase 2a, Ascending Dose, Placebo-Controlled Study to Evaluate the Safety of CTX-100 (Formerly ETX-100) Inhalation Solution in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Safety Study of CTX-100 Inhalation Solution (Formerly ETX-100)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Turino, Gerard, M.D. (Individual)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: C100-005; 1R01HL081489-01A1 (NIH)
Record Dates: First submitted 2009-09-22; First posted 2009-10-12 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0.01% CTX-100 (formerly ETX-100) (Active Comparator)
  Interventions: Drug: CTX-100 (formerly ETX-100) (hyaluronic acid)
- 0.03% CTX-100 (formerly ETX-100) (Active Comparator)
  Interventions: Drug: CTX-100 (formerly ETX-100) (hyaluronic acid)
- Placebo (Placebo Comparator)
  Interventions: Drug: CTX-100 (formerly ETX-100) (hyaluronic acid)

INTERVENTIONS:
Drug: CTX-100 (formerly ETX-100) (hyaluronic acid) — 3 mL of either 0.01%, 0.03% CTX-100 (formerly ETX-100), or placebo will be dispensed into the PARI LC STAR nebulizer and inhaled using the PARI Ultra II compressors.
  Number of cycles: if the study drug (0.01% CTX-100 Inhalation Solution or placebo) bid is well tolerated in the first cohort, the second cohort of subjects will begin dosing with 0.03% CTX-100 Inhalation Solution or placebo in the same manner as the first cohort.
  Other Names: CTX-100; ETX-100; Hyaluronic acid

SUMMARY:
The purpose of the study is to evaluate the safety of administering repeated doses of CTX-100 (formerly ETX-100) to subjects with smoking-related chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
The study primarily aims to establish safety and evaluate biochemical activity of CTX-100 (formerly ETX-100) with respect to elastin breakdown, but will also concurrently gather data that may point to efficacy. The preliminary efficacy results will be used to assist in the design of subsequent phase 2b clinical studies of longer duration to examine both efficacy and safety of CTX-100 as a therapy for chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent and comply with study requirements.
* Men or women aged 40 through 75 years at the time of consent.
* At least 10-pack years (average packs/day x number of years) of cigarette use, and either current smoker or ex-smoker.
* Diagnosis of COPD at screening consistent with National Institutes of Health guidelines.
* Evidence of emphysema on chest x-ray.
* A ratio of prebronchodilator FEV1 to forced vital capacity (FVC) of ≤ 70% at screening.
* FEV1 ≥ 50% (prebronchodilator) and ≤ 79% (postbronchodilator) of predicted normal at screening.
* Clinical laboratory tests (complete blood count, serum chemistry, and urinalysis) within normal limits or clinically acceptable to the PI/sponsor at screening.
* Women of childbearing potential and men who are sexually active must agree to use an adequate method of contraception (oral contraceptives, depot progesterone, condom plus spermicide, or IUD) during the study and for 1 month after the final dose of study drug.

Exclusion Criteria:

* Subjects with a measured DLCO of ≤ 50%, or unable to perform a reproducible DLCO.
* Subjects unable to perform 3 reproducible spirometry tests after 5 attempts.
* Upper or lower respiratory tract infection within 2 weeks prior to screening and baseline (day 1).
* Presence of clinically relevant abnormality on chest x-ray (other than evidence of emphysema) at screening or within the previous 12 months.
* Use of supplemental oxygen therapy.
* Requirement for ventilatory support within the last year.
* Exacerbation requiring treatment with systemic corticosteroids within the last 3 months.
* History of lung transplant.
* Presence of clinically relevant abnormality on electrocardiogram (ECG).
* Any medical condition that, in the investigator's judgment, would compromise study participation or the evaluation of the study drug.
* Women who are pregnant or breastfeeding.
* Receipt of an investigational drug within 30 days prior to screening (including subjects who participated in the first phase of this study).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Assessment of vital signs, laboratory tests, carbon monoxide (CO) diffusing capacity, oxygen saturation, electrocardiograms (ECGs), physical examinations, and adverse events | 1 month

SECONDARY OUTCOMES:
Assessment of elastin breakdown as measured by levels of elastin crosslinking amino acids desmosine/isodesmosine (D/I) in induced sputum, plasma, and urine. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Turino, M.D., Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (3):
- United States (3):
  - Arizona Research Associates, Tucson, Arizona
  - VA Harbor Medical Center, New York, New York
  - St. Luke's-Roosevelt Hospital Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes